CLINICAL TRIAL: NCT06136351
Title: A Study of the Zanubrutinib Given in Combination With Bendamustine and Rituximab in (Elderly or TP53 Alterations or Chemotherapy Intolerance) Patients With Newly Diagnosed Mantle Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZBR-01
Record Dates: First submitted 2023-09-25; First posted 2023-11-18 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Lymphoma, Mantle-Cell
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — zanubrutinib; Rituximab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZBR (Experimental)
  Interventions: Drug: Zanubrutinib; Drug: Rituximab; Drug: Bendamustin

INTERVENTIONS:
Drug: Zanubrutinib — 160 mg bid po, until disease progression, intolerance of drug toxicity or death, otherwise maintaining during the 2 years of follow-up
Drug: Rituximab — 375 mg/m^2 ivgtt, D0 of each 28-day cycle
Drug: Bendamustin — 90mg/m^2 ivgtt, D0 of each 28-day cycle

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Zanubrutinib given in combination with bendamustine and rituximab in (elderly or TP53 alterations or chemotherapy intolerance) patients with newly diagnosed mantle cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* 18 years

  * Histopathologically confirmed mantle cell lymphoma according to the 5th edition of the World Health Organization (WHO)
  * FISH with del(17p)/TP53 mutation or ≥65 years; or<65 years but chemotherapy intolerance;
  * Life expectancy of > 3 months (in the opinion of the investigator);
  * Creatinine Clearance Rate (CCR) ≥ 50 mL/min or estimated Glomerular Filtration ●Rate (eGFR) ≥ 60 mL/(min·1.73 m^2);
  * International Normalized Ratio (INR) ≤ 1.5 and activated Partial Thromboplastin Time (aPTT) ≤ 1.5 times the upper limit of normal;
  * Left Ventricular Ejection Fraction (LVEF) ≥ 50%;
  * Agreeing to provide written informed consent prior to any special examination or procedure for the research on their own or legal representative.

Exclusion Criteria:

* Pregnant or lactating women;
* Known Hepatitis B Virus (HBV) and/or Hepatitis C Virus (HCV) infection (HBV infection refers to HBV-DNA > detectable limit);
* With acquired or congenital immunodeficiency;
* With congestive heart failure in 6 months before enrollment, New York Heart Association (NYHA) heart function class III or IV, or LVEF < 50%;
* Known to be allergic to the test drug ingredients;
* Diagnosed with or being treated for malignancy other than lymphoma;
* With severe infection;
* Substance abuse, medical, psychological, or social conditions that may interfere with the subjects' participation in the study or evaluation of the study results;
* Deemed unsuitable for the group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
2-year Progression-Free Survival | 2 years
  Progression-free survival was defined as the time from the date of first treatment until the date of the first documented day of disease progression or relapse, according to 2014 Lugano criteria, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
ORR | End of treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=28 days]
  Objective Remission Rate (ORR) is defined as the proportion of patients with complete remission (CR) and partial remission (PR)
CRR | End of treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=28 days]
  Complete Remission Rate (CRR) is defined as the proportion of patients with CR
OS | Baseline up to data cut-off (up to approximately 2 years)
  Overall survival (OS) refers to the time from receiving the first dose to death from any cause
Adverse Events | Baseline up to data cut-off (up to approximately 2 years)
  Any harmful reaction that occurs during the treatment of a disease according to the normal usage and dosage of a drug, which is unrelated to the purpose of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No